CLINICAL TRIAL: NCT03294603
Title: A Phase 1, Single-center, Open-label Study to Evaluate the Metabolism and Excretion of (14C)-CC-220 in Healthy Male Subjects
Brief Title: Radiolabeled Study of CC-220 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC-220-CP-006; U1111-1202-3955 (Registry Identifier: WHO)
Record Dates: First submitted 2017-09-22; First posted 2017-09-27 (Actual); Last update posted 2017-10-25 (Actual); Status verified 2017-10

CONDITIONS: Healthy Volunteer
Keywords: Healthy Volunteer; CC-220; Male
MeSH Terms: interventions — iberdomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [14C]-CC-220 solution (Experimental): A single oral dose of 1 mg [14C]-CC-220 solution, containing approximately 1.4 μCi of radioactivity, will be administered on Day 1 under fasted conditions.
  Interventions: Drug: CC-220; Radiation: [14C]

INTERVENTIONS:
Drug: CC-220 — 1mg [14C]-CC-220 will be administered as a single dose
Radiation: [14C] — Single dose of [14C]-CC-220 will contain approximately 1.4 μCi of radioactivity

SUMMARY:
This is a single-center, open-label study to characterize the biotransformation and excretion of [14C]-CC-220 in healthy male subjects. Each subject will participate in screening, a treatment phase (including baseline), and a follow-up phone call. Subjects will be screened for eligibility. Subjects who have met all inclusion criteria and none of the exclusion criteria at screening will return to the study site on Day -1, and will be domiciled at the study site from Day -1 to Day 10. On Day 1, subjects will receive a single oral dose of 1 mg [14C]-CC-220 under fasted conditions. Blood, urine, and fecal samples will be collected throughout the study for pharmacokinetic (PK; inclusive of metabolite profiling / characterization), mass balance, and/or clinical laboratory assessments. Safety will be monitored throughout the study. Subjects will be discharged from the study site on Day 10 following completion of the scheduled study procedures and satisfactory safety review. Subjects will participate in a follow-up phone call within 5 to 7 days following discharge.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is ≥ 18 and ≤ 55 years of age at the time of signing the informed consent form (ICF).
2. Subject is male.
3. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
4. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
5. Subject is in good health, as determined by the Investigator based on a physical examination at screening.
6. Subject agrees to abide by the requirements and restrictions outlined in the CC-220 Pregnancy Prevention Plan for Subjects in Clinical Trials.
7. Subject must agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or a female of childbearing potential (FCBP)1 while participating in the study and for at least 90 days following administration of CC-220, even if he has undergone a successful vasectomy.
8. Subject has a body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
9. Subject has clinical laboratory safety test results that are within normal limits or considered not clinically significant by the Investigator. Platelet count, absolute neutrophil count (ANC), and absolute lymphocyte count (ALC) must be above the lower limit of normal at screening.
10. Subject is afebrile, with supine systolic blood pressure (BP) ≥ 90 and ≤ 140 mmHg, supine diastolic BP ≥ 50 and ≤ 90 mmHg, and pulse rate ≥ 40 and ≤ 110 bpm at screening.
11. Subject has a normal or clinically acceptable 12-lead electrocardiogram (ECG), with a QTcF value ≤ 430 msec, at screening.

Exclusion Criteria:

1. Subject has any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subject was exposed to an investigational drug (new chemical entity) within 30 days prior to dosing, or 5 half-lives of that investigational drug, if known (whichever is longer).
5. Subject has used any prescribed systemic or topical medication (including but not limited to analgesics, anesthetics, etc) within 14 days or 5 half-lives of that medication, whichever is longer, prior to dosing.
6. Subject has used any non-prescribed systemic or topical medication (including vitamin/mineral supplements and herbal medicines) within 7 days prior to dosing.
7. Subject has used CYP3A inducers and/or inhibitors (including St. John's Wort) within 30 days prior to dosing. The Indiana University "Cytochrome P450 Drug Interaction Table" should be utilized to determine inducers and/or inhibitors of CYP3A.
8. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, eg, bariatric procedure.

   Note: prior appendectomy is acceptable, but prior cholecystectomy would result in exclusion from the study.
9. Subject donated blood or plasma within 8 weeks prior to dosing to a blood bank or blood donation center.
10. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years prior to dosing, or positive drug test reflecting consumption of illicit drugs.
11. Subject has a history of alcohol abuse (as defined by the current version of the DSM) within 2 years prior to dosing, or positive alcohol test.
12. Subject is known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.
13. Subject smokes > 10 cigarettes per day, or equivalent in other tobacco products (self-reported).
14. Subject has received immunization with a live or live attenuated vaccine within 2 months prior to dosing or is planning to receive immunization with a live or live attenuated vaccine for 2 months following dosing.
15. Subject participated in a radiolabeled drug study, where exposures are known to the Investigator, within the previous 4 months prior to check-in (Day -1); or participated in a radiolabeled drug study, where exposures are not known to the Investigator, within the previous 6 months prior to check-in (Day -1). The total 12-month exposure from this study and a maximum of 2 other previous studies within 4 to 12 months of this study will be within the CFR recommended levels considered safe, per US Title 21 CFR 361.1: less than 5,000 mrem whole body annual exposure, with consideration given to the half-lives of the previous radiolabeled study drugs received.
16. Subject was exposed to significant radiation (eg, serial X-ray or computed tomography scans, barium meal, current employment in a job requiring radiation exposure monitoring) within 12 months prior to check-in (Day -1).
17. History of less than 1 to 2 bowel movements per day.
18. Subject is part of the study site personnel or a family member of the study site staff.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2017-09-11 (Actual); Primary Completion 2017-10-16 (Actual); Study Completion 2017-10-16 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics -Total [14C]-Radioactivity (RA) | Up to approximately Day 10
  Total [14C]-RA in whole blood, plasma, urine, and feces (and vomit, if applicable) will be measured via AMS.
Pharmacokinetics - Cumulative excretion of total [14C]-RA | Up to approximately Day 10
  Total RA recovery will be computed as the sum of the cumulative excretion (as % dose) in urine and feces (and vomit, if applicable).
Pharmacokinetics - Total [14C]-RA whole blood-to-plasma | Up to approximately Day 10
  Total [14C]-RA in whole blood and plasma will be converted to ngEq/mL concentration of [14C]-CC-220 based on specific activity of the dose.
Pharmacokinetics - metabolite profiling/characterization | Up to approximately Day 10
  Percentage of the administered dose attributed to CC-220 and metabolite(s), and the RA of [14C]-CC-220 and metabolite(s), as appropriate, will be estimated.
Pharmacokinetics -Cmax | Up to approximately Day 10
  Observed maximum plasma concentration, provided sufficient data available
Pharmacokinetics -AUC | Up to approximately Day 10
  Area under the concentration-time curve, provided sufficient data available
Pharmacokinetics -Tmax | Up to approximately Day 10
  Time to Cmax, provided sufficient data available
Pharmacokinetics -t1/2 | Up to approximately Day 10
  Terminal elimination half-life, provided sufficient data available

SECONDARY OUTCOMES:
Adverse Events (AEs) | From enrollment until at least 28 days after completion of study treatment
  Number of participants with adverse event

CONTACTS AND LOCATIONS:
Overall Officials: Maria Palmisano, MD, Study Director — Celgene
Locations (1):
- Covance Clinical Research Unit, Madison, Wisconsin, United States

REFERENCES:
- [Derived] Cheng Y, Wang X, Liu L, Silva J, Thomas M, Li Y. A Phase I, Open-Label, Mass Balance Study of [14C]-Iberdomide in Healthy Subjects. Eur J Drug Metab Pharmacokinet. 2024 May;49(3):355-365. doi: 10.1007/s13318-024-00886-4. Epub 2024 Mar 23. PMID 38521893